CLINICAL TRIAL: NCT05377372
Title: Early Life Exposures Among Children With Sickle Cell Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Brandi Pernell, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300003639; 5K23HL159280 (NIH)
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease; Adverse Childhood Experiences; Breastfeeding
Keywords: Sickle cell disease; Adverse Childhood Experiences; Breastfeeding
MeSH Terms: conditions — Anemia, Sickle Cell; Breast Feeding | interventions — Observation

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding Intervention Group (Experimental): Ten mother-infant dyads will be recruited to a six-month, community-based intervention aimed to promote sustained breastfeeding for at least six months among mothers of infants with sickle cell disease. The intervention will include an online, social media-based support group, online educational modules, monthly in-person educational sessions, access to free breast pump rentals, and monthly peer-led home visits by certified Vanderbilt-affiliated Maternal Infant Health Outreach Specialists. We obtain whole blood specimens for analysis of oxidative stress and inflammation at 3, 6, 12 and 24 months.
  Interventions: Behavioral: Breastfeeding support group
- Observation Group (Other): A 24 month observation of 10 mother-infant dyads affected by sickle cell disease that initiate breastfeeding. These dyads will observed for breastfeeding exclusivity/dosage and duration. We obtain whole blood specimens for analysis of oxidative stress and inflammation at 3, 6, 12 and 24 months.
  Interventions: Other: Observation

INTERVENTIONS:
Behavioral: Breastfeeding support group — community-based breastfeeding support group aimed to increase exclusive breastfeeding success rates among Black women
  Arms: Breastfeeding Intervention Group
Other: Observation — Observe prospectively for breastfeeding initiation, duration and longitudinal health of child with sickle cell disease
  Arms: Observation Group

SUMMARY:
This study is being conducted to determine the relationship between early childhood exposures, such as Adverse Childhood Experiences, Social Determinants of Health and nutrition/breastfeeding, among children with sickle cell disease, and behavioral interventions aimed to reshape psychological resilience and lifestyle factors towards positive health outcomes.

DETAILED DESCRIPTION:
During year 3 of the award period, 20 mother-infant dyads will be randomly assigned to either a community-based breastfeeding support group or observation. Acceptability to enrollment, intervention adherence for at least 6 months and preliminary effectiveness will be captured. Biomarkers of inflammation, development of asthma and incidences of pain and/or acute chest syndrome will be compared among the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* mother of infant with sickle cell disease
* resides within the city of Birmingham, Alabama or in close proximity

Exclusion Criteria:

* prescribed teratogenic medications
* no/limited internet access

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptance and Retention of Mothers of Infants with Sickle Cell Disease to a Community-based Breastfeeding Intervention | 6 months
  acceptance (number of mothers enrolled/number of mothers approached) and retention (number of mothers to complete 6 month support group intervention/number enrolled)
Preliminary Effectiveness | 2 years
  Percentage of mothers of infants with sickle cell disease that successful complete 6 months of breastfeeding, comparing the intervention vs. control groups

SECONDARY OUTCOMES:
Asthma | 4 year follow up period
  Prevalence of asthma among children with sickle cell disease that were breastfed compared to those that were not
Acute chest syndrome | 4 year follow up period
  Incidence rate of episodes of acute chest syndrome among children with sickle cell disease that were vs. were not breastfed

CONTACTS AND LOCATIONS:
Overall Officials: Brandi M Pernell, DNP, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
I will share by IPD. I do not have a URL at this time and could not get my application to submit without submitting a URL